CLINICAL TRIAL: NCT03019822
Title: Role of Dopamine, Serotonin and 5-HT2A Receptors in Emotion Processing
Acronym: LAM
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: BASEC 2016-01827
Record Dates: First submitted 2016-12-22; First posted 2017-01-13 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Healthy
MeSH Terms: interventions — Lysergic Acid Diethylamide; N-Methyl-3,4-methylenedioxyamphetamine; Amphetamine; Dextroamphetamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo, LSD, d-Amphetamine, MDMA (Other): Cross-over within-subjects design with all treatment conditions, arms starting with either Placebo, lysergic acid diethylamide (LSD), d-Amphetamine or methylenedioxymethamphetamine (MDMA) and followed by all other drugs each separated by a wash-out phase
  Interventions: Drug: LSD; Drug: MDMA; Drug: Amphetamine; Drug: Placebo
- LSD, d-Amphetamine, MDMA, Placebo (Other): Cross-over within-subjects design with all treatment conditions, arms starting with either Placebo, LSD, d-Amphetamine or MDMA and followed by all other drugs each separated by a wash-out phase
  Interventions: Drug: LSD; Drug: MDMA; Drug: Amphetamine; Drug: Placebo
- d-Amphetamine, MDMA, LSD, Placebo (Other): Cross-over within-subjects design with all treatment conditions, arms starting with either Placebo, LSD, d-Amphetamine or MDMA and followed by all other drugs each separated by a wash-out phase
  Interventions: Drug: LSD; Drug: MDMA; Drug: Amphetamine; Drug: Placebo
- MDMA, LSD, Placebo, d-Amphetamine,, (Other): Cross-over within-subjects design with all treatment conditions, arms starting with either Placebo, LSD, d-Amphetamine or MDMA and followed by all other drugs each separated by a wash-out phase
  Interventions: Drug: LSD; Drug: MDMA; Drug: Amphetamine; Drug: Placebo

INTERVENTIONS:
Drug: LSD — 100ug per os, single dose
  Other Names: Lysergic Acid Diethylamide
Drug: MDMA — 125mg per os, single dose
  Other Names: 3,4-methylenedioxymethamphetamine
Drug: Amphetamine — 40.3mg per os, single dose
  Other Names: d-amphetamine sulfate
Drug: Placebo — Capsules containing mannitol looking identical to the other drugs

SUMMARY:
The study will test the effect of dopamine, serotonin, and direct 5-HT2A receptor stimulation on empathy, mood perception, and amygdala activity to fearful stimuli. In addition, we predict associations between subjective effects/alterations in emotion processing tests and functional imaging (fMRI) activity.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 25 and 50 years.
2. Sufficient understanding of the German language
3. Subjects understand the procedures and the risks associated with the study.
4. Participants must be willing to adhere to the protocol and sign the consent form.
5. Participants must be willing to refrain from taking illicit psychoactive substances during the study.
6. Participants must be willing to drink only alcohol-free liquids and no coffee, black or green tea, or energy drink after midnight of the evening before the study session, as well as during the study day.
7. Participants must be willing not to drive a traffic vehicle or to operate machines within 48 h after substance administration.
8. Women of childbearing potential must have a negative pregnancy test at the beginning of the study. Pregnancy tests are repeated before each study session. Women and men must agree to use an effective form of birth control (double-barrier method).
9. Body mass index 18-29 kg/m2.

Exclusion Criteria:

1. Chronic or acute medical condition
2. Hypertension (>140/90 mmHg) or Hypotension (SBP<85 mmHg)
3. Current or previous major psychiatric disorder
4. Psychotic disorder in first-degree relatives
5. Illicit substance use (with the exception of cannabis) more than 10 times or any time within the previous two months.
6. Pregnant or nursing women.
7. Participation in another clinical trial (currently or within the last 30 days)
8. Use of medications that may interfere with the effects of the study medications (any psychiatric medications).
9. fMRI related criteria including: metal implants (clips from operations, cochlea, large red/yellow tattoos in the neck area)
10. Tobacco smoking (>10 cigarettes/day)
11. Consumption of alcoholic drinks (>10/week)

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-08-11 (Actual); Study Completion 2018-09-04 (Actual)

PRIMARY OUTCOMES:
Emotional enhancement as determined by fMRI | 12 hours
  Emotional enhancement (empathy, oxytocin, mood perception, fMRI amygdala blood oxygen level-dependent (BOLD) signal reactivity to fearful stimuli)
fMRI brain activity | 1 hour
  Associations between subjective effects/alterations in emotion processing with fMRI amygdala BOLD activity

SECONDARY OUTCOMES:
Resting State fMRI | 1 hour
  Association between emotional enhancement and resting state fMRI neuronal activity
Effect Modulation by personality traits (assessed with questionnaires), | 12 hours
  Effect modulation by personality traits (assessed with questionnaires), baseline amygdala reactivity to fear in the fMRI, and genetic polymorphisms determined by genotyping of each subject
Effect Modulation by amygdala reactivity to fear (assessed in the fMRI) | 12 hours
  Effect modulation by personality traits (assessed with questionnaires), baseline amygdala reactivity to fear in the fMRI, and genetic polymorphisms determined by genotyping of each subject
Effect Modulation by genetic polymorphisms (determined by genotyping of each subject) | 12 hours
  Effect modulation by personality traits (assessed with questionnaires), baseline amygdala reactivity to fear in the fMRI, and genetic polymorphisms determined by genotyping of each subject

CONTACTS AND LOCATIONS:
Overall Officials: Matthias E Liechti, MD, MAS, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided